CLINICAL TRIAL: NCT02862236
Title: The Acute Effect of Hypericum Perforatum on Short-Term Memory in Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prof. Eldad Yechiam (Other)
Collaborators: Beer Yaakov - Ness Ziona Mental Health Center (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Eldad Yechiam, Associate Professor, Behavioral Science, Technion, Israel Institute of Technology
Organization: Technion, Israel Institute of Technology (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-2016
Record Dates: First submitted 2016-07-25; First posted 2016-08-10 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Subclinical Anxious Adults; Nootropic Potential of Hypericum and Alprazolam; Healthy Adults
MeSH Terms: interventions — Hypericum extract LI 160

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypericum perforatum (Remotiv, 250 mg) (Experimental)
  Interventions: Drug: Hypericum perforatum extract
- Hypericum perforatum (Remotiv, 500 mg) (Experimental)
  Interventions: Drug: Hypericum perforatum extract

INTERVENTIONS:
Drug: Hypericum perforatum extract — 250 or 500 mg Remotiv capsules of hypericum perforatum extract, p.o.

SUMMARY:
Rationale Over-the-counter drugs containing hypericum perforatum (H. perforatum), have been argued to improve memory and sustained attention. So far, these claims have not been supported in human studies. However, previous studies used rather high dosages, and little is known about the acute effect of small dosages.

Objective We evaluated whether an acute treatment with Remotiv 500 and Remotiv 250 (500 or 250 mg of H. perforatum quantified to either 1 or 0.5 mg of hypericin) improved memory, sustained attention, as well as mood and state anxiety in healthy adults.

Method A single dosage, randomized, double blind, placebo-controlled trial was conducted with 82 student participants (33 women). Each participant received placebo in one session and one of two dosages in the other session. Order of the sessions and dosage conditions were randomized between subjects. Participants completed a battery of tasks assessing short-term memory capacity and sustained attention.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults 18 to 40 years old.

Exclusion Criteria:

* 1. Demographics: Under 18 years of age or older than 40; pregnant or nursing women; non-fluent Hebrew speakers.

  2. Body weight: less than 50 kg and more than 90 kg (to ensure effective drug dosage).

  3. Mental health: Diagnosed with any DSM-V disorder (including ADHD, learning disabilities). These DSM-V disorders may be included in the research: sexual dysfunctions, sleeping disorders and mild-moderate anxiety disorders.

  4. Any motor disability hampering a participant's ability to perform the experimental task.

  5. Consumption of any psychoactive substance within the last 72 hours. 6. Ongoing medical problems or use of any substances (e.g., other prescribed medications) which may interact negatively with any of the three drugs used in the experiment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Go/no-go task | one-two hours after drug administration
  A computerized cognitive task: aimed to measure attention and impulsivity: errors of omission and commission
Digit span task | one-two hours after drug administration
  A computerized cognitive task; accuracy of recalling
Symmetry span task | one-two hours after drug administration
  A computerized cognitive task; accuracy of responses
Operation span task | one-two hours after drug administration
  A computerized cognitive task; accuracy of responses
Groton's Maze task | one-two hours after drug administration
  A computerized task

SECONDARY OUTCOMES:
DASS-21 | one-two hours after drug administration
  A self-report questionnaire; scoring of relevant state anxiety items
PANAS | one-two hours after drug administration
  A self-report questionnaire
STAI | one-two hours after drug administration
  A self-report questionnaire; scoring of relevant state anxiety items

CONTACTS AND LOCATIONS:
Overall Officials: Mili Bar-Shaked, MD, Principal Investigator — Beer Yaakov - Ness Ziona Mental Health Center; Eldad Yechiam, PhD, Study Director — Technion, Israel Institute of Technology
Locations (1):
- Technion, Israel Institute of Technology, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yechiam E, Ben-Eliezer D, Ashby NJS, Bar-Shaked M. The acute effect of Hypericum perforatum on short-term memory in healthy adults. Psychopharmacology (Berl). 2019 Feb;236(2):613-623. doi: 10.1007/s00213-018-5088-0. Epub 2018 Oct 31. PMID 30382352